CLINICAL TRIAL: NCT05935865
Title: Monitoring of the Influence of Approved PH-therapies RV-PA Coupling
Status: Recruiting | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Other Study IDs: 211/22
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Pulmonary Hypertension
Keywords: Monitoring; RV-PA Coupling; Pulmonary Hypertension; Right Ventricle
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the acute (days) changes in right ventricular functions caused by initiation of pharmacological therapies in patients with precapillary pulmonary hypertension. The main question it aims to answer is:

• Course of afterload and intrinsic contractility throughout the hospital stay Participants will be equipped with a device for continuous monitoring and recording of the right ventricular pressure signal.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) arises as a result of a vascular pathology affecting the pulmonary vessels, leading to an increase in resistance within the pulmonary circulation. The ability of the right ventricle to adapt to the elevated pressures caused by increased afterload is crucial for the progression and symptoms of the disease. This adaptation of the right ventricle to its afterload is referred to as ventriculoarterial coupling or RV-PA coupling, described by the ratio of contractility to afterload. Invasive pressure-volume loops (PV loops) are the gold standard for assessing RV-PA coupling. The loss of RV-PA coupling is considered a crucial factor in the development of right heart failure, the leading cause of mortality in patients with pulmonary hypertension. Therefore, reliable assessment of right cardiac function is essential for physicians to make informed decisions regarding further invasive diagnostics or therapy adjustments. Approved medications for the treatment of pulmonary arterial hypertension primarily induce pulmonary vasodilation, leading to a reduction in right ventricular afterload. The effects on right ventricular contractility and function, as represented by RV-PA coupling, are currently poorly understood and may not be consistent. In this study, 100 patients with PH requiring an inpatient stay for right heart catheterization will be equipped with a mobile, wireless system for invasive measurement of right ventricular pressure - the CorLog system (emka MEDICAL, Aschaffenburg, Germany). By combining continuously recorded pressure profiles with 3D echocardiographic volumetry, we will be able to generate PV loops and assess RV-PA coupling at various time points. The continuous monitoring of right ventricular pressure profiles throughout the entire hospital stay will allow us to capture the effects of newly initiated or expanded pulmonary vascular therapy on RV-PA coupling not only immediately but over several days. Furthermore, the 3D echocardiographic datasets will be analyzed using specialized software (ReVISION®, Argus Cognitive, Inc, Lebanon, NH) to mechanistically quantify the right ventricular contraction pattern and capture the immediate impact of pulmonary vasoreactive therapy on it. Additionally, a data pool will be created to validate the calculation of ejection fraction and RV-PA coupling based solely on pressure signals.

ELIGIBILITY:
Inclusion Criteria:

* Initial diagnosis of PH (treatment-naive incident PH) of the Nice classifications 1 (PAH), 3 (PH related to lung diseases/hypoxia), and 4 (CTEPH), or known PH under ongoing vasoreactive therapy
* No contraindications for right heart catheterization, conductance catheterization, or CorLog implantation
* Written consent from the patient or their legal guardian

Exclusion Criteria:

* Absence of written consent
* Invasive exclusion of PH
* Age < 18 years
* Presence of contraindications for right heart catheterization, conductance catheterization, or CorLog implantation
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with pre-capillary pulmonary hypertension (Nice classification groups 1, 3, or 4) who are scheduled to undergo right heart catheterization for clinical reasons as part of invasive diagnostics for:
  1. Establishing a diagnosis when there is a non-invasive suspicion of pulmonary hypertension.
  2. Performing invasive hemodynamic assessment in patients already receiving vasoactive therapy, with the question of therapy escalation, particularly in cases of right cardiac decompensation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2025-02-13 (Estimated); Study Completion 2026-02-13 (Estimated)

PRIMARY OUTCOMES:
Afterload | 3-7days
  Responce of afterload (calculated from PV loops [Ea]) afterload during hospitalization to the initiation or escalation of pulmonary vascular therapy
Contractility | 3-7days
  Response of contractility (calculated from PV loops [Ees]) during hospitalization to the initiation or escalation of pulmonary vascular therapy
Coupling | 3-7days
  Response of Coupling (calculated from PV loops [Ees/Ea]) during hospitalization to the initiation or escalation of pulmonary vascular therapy
Validation of Echo/CorLog PV-Loops | On first day
  Validation of Echo/Corlog-generated PV loops based on conductance catheter-generated PV loops

SECONDARY OUTCOMES:
Validation of pressure-only methods | 3-7days
  Validation of methods for calculating ejection fraction and RV-PA coupling using ventricular pressure signals
Contraction patterns | 3-7 days
  Analysis of volumetric datasets of the right ventricle using ReVISION software. Isolated quantification of right ventricular systolic shortening along the ventricular axes in 3-dimensional space.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Justus Liebig University Giessen, Universities of Giessen and Marburg Lung Center (UGMLC), German Center for Lung Research (DZL), Giessen, Hesse, Germany